CLINICAL TRIAL: NCT01495052
Title: Effect of Organic Naked Oat With Whole Germ on Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Li (Other)
Responsible Party: Sponsor-Investigator, Yong Li, Professor, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ONOG-0001; ONOG-0001-01 (Other: Beijing Nutrition society)
Record Dates: First submitted 2011-12-09; First posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes Mellitus
Keywords: naked oat (Avena nuda L.); diabetes mellitus; RCT
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual care group (No Intervention): The usual care group was used as control group and didn't receive any intervention except standard health advice at the beginning and the end of the study.
- diet group (No Intervention): This group received systematic education about nutrition and diabetes combined with a structured dietary intervention.
- 50g-ONOG plus diet group (Experimental): This group received systematic education about nutrition and diabetes combined with a structured dietary intervention. Participants in the 50g-ONOG plus diet groups were asked to replace their customarily used staple food with oat porridge containing 50g ONOG.
  Interventions: Dietary Supplement: organic naked oat with whole germ (ONOG)
- 100g-ONOG plus diet group (Experimental): This group received systematic education about nutrition and diabetes combined with a structured dietary intervention. Participants in the 100g-ONOG plus diet groups were asked to replace their customarily used staple food with oat porridge containing 100g ONOG.
  Interventions: Dietary Supplement: organic naked oat with whole germ (ONOG)

INTERVENTIONS:
Dietary Supplement: organic naked oat with whole germ (ONOG) — The experimental product was ONOG (Inner Mongolia Sanzhuliang Natural Oats Industry Corporation), which was produced in the northwest part of China, applying with the organic standards. Participants in the 50g and 100g-ONOG plus diet groups were asked to replace their customarily used staple food with oat porridge containing 50g or 100g ONOG.
  Other Names: organic naked oat with whole germ (ONOG),
  Arms: 100g-ONOG plus diet group; 50g-ONOG plus diet group

SUMMARY:
Dietary modification is of great essential for the prevention and treatment of type 2 diabetes mellitus. Common oat (Avena sativa L.) and its products showed a great potential benefits on NCDs including type 2 diabetes mellitus. But data about such effects of naked oat (Avena nuda L.) is still unavailable. The investigators aimed to examine the effects of organic naked oat with whole germ (ONOG) plus diet on patients with type 2 diabetes.

After a pre-study with healthy adults, a randomized, single-blinded, multi-arm parallel trial of 30 days would be carried out in adults of 50-65 years old with type 2 diabetes. Participants would be randomly assigned to one of the four following groups: usual care group (only basic health advice, no other interventions), diet group (systematic education, structured dietary), 50g-ONOG plus diet group (all the interventions of diet group plus replacement of 50g ONOG per day) and 100g-ONOG plus diet group. A regular follow-up for years would be carried out to predict the long-term effects of ONOG plus diet intervention on patients with type 2 diabetes.

The investigators hypothesized that ONOG combined with diet would have better effects on glycaemia and insulin resistance control in addition to those yielded by diet or usual care.

ELIGIBILITY:
Inclusion Criteria:

* all adults aged 50-65 years old with Type 2 Diabetes Mellitus
* stable physical condition
* fasting plasma glucose (FPG) concentration ≥7.8mmol/L or 2-h postprandial blood glucose (PG) ≥11.1mmol/L after 75g oral dextrose with an glycated hemoglobin (HbA1c)>7 %, stable medication.

Exclusion Criteria:

* pregnancy
* breastfeeding
* severe renal or hepatic complications
* treatment by glucocorticoid
* having pancreatic disease or malignancy in recent 3 months
* other factors that may limit adherence to interventions or affect conduct of the trial or participation in another supplementary feeding programme.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
change from baseline in Hb1Ac concentration Hematology index detection Hematology index detection Hematology index detection Hematology index detection Hematology index detection | baseline, 30 days, 6 months and 1 year
  Venous blood samples were collected for determination of glycosylated haemoglobin (HbA1c).Changes in outcomes were calculated as values at the end of the intervention period minus those of baseline.
changes from baseline in insulin resistance Hematology index detection Hematology index detection Hematology index detection Hematology index detection Hematology index detection | baseline, 30 days, 6 months and 1 year
  Venous blood samples were collected for determination of serum insulin.Insulin resistance was measured by HOMO-IR, calculated with the following formula:
  HOMO-IR=Fasting serum insulin(μU/mL)*FPG(mmol/L)/22.5

SECONDARY OUTCOMES:
changs from baseline in plasma glucose | baseline, 30 days, 6 months and 1 year
  Venous blood samples were collected for determination of fasting plasma glucose(FPG), postprandial blood glucose (PG).Changes in outcomes were calculated as values at the end of the intervention period minus those of baseline.
changes from baseline in lipid profile | baseline, 30 days, 6 months and 1 year
  Venous blood samples were collected for determination of total triglycerides (TG), total cholesterol (TC), low-density lipoprotein cholesterol (LDL-c), high-density lipoprotein cholesterol (HDL-c). Changes in outcomes were calculated as values at the end of the intervention period minus those of baseline.
changes from baseline in BMI | baseline, 30 days, 6 months and 1 year
  Weight and height were measured at each time. BMI was calculated as weight divided by square height.Changes in outcomes were calculated as values at the end of the intervention period minus those of baseline.
changes from baseline in plasma levels of total glutathione peroxidase, malondialdehyde(MDA), superoxide dismutase (SOD), IL-6 and TNF-а | baseline and 30 days
  Venous blood samples were collected for determination of total glutathione peroxidase, malondialdehyde(MDA), superoxide dismutase (SOD), IL-6 and TNF-а. Changes in outcomes were calculated as values at the end of the intervention period minus those of baseline.
changes from baseline in WHR | baseline, 30 days, 6 months and 1 year
  waist circumference and hip circumference were measured at each time. WHR was calculated as waist circumference divided by hip circumference.Changes in outcomes were calculated as values at the end of the intervention period minus those of baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Arms Industry New Century Hotel, Baotou, Inner Mongolia, China

REFERENCES:
- [Derived] Li X, Cai X, Ma X, Jing L, Gu J, Bao L, Li J, Xu M, Zhang Z, Li Y. Short- and Long-Term Effects of Wholegrain Oat Intake on Weight Management and Glucolipid Metabolism in Overweight Type-2 Diabetics: A Randomized Control Trial. Nutrients. 2016 Sep 7;8(9):549. doi: 10.3390/nu8090549. PMID 27618090
- [Derived] Gu J, Jing L, Ma X, Zhang Z, Xu M, Wang J, Li Y. Naked oat combined with a structured dietary intervention affects oxidative stress but not inflammation in diabetic dyslipidemia. Nutr Metab Cardiovasc Dis. 2014 Dec;24(12):e35-7. doi: 10.1016/j.numecd.2014.08.009. Epub 2014 Sep 16. No abstract available. PMID 25315670
- [Derived] Ma X, Gu J, Zhang Z, Jing L, Xu M, Dai X, Jiang Y, Li Y, Bao L, Cai X, Ding Y, Wang J, Li Y, Li Y. Effects of Avena nuda L. on metabolic control and cardiovascular disease risk among Chinese patients with diabetes and meeting metabolic syndrome criteria: secondary analysis of a randomized clinical trial. Eur J Clin Nutr. 2013 Dec;67(12):1291-7. doi: 10.1038/ejcn.2013.201. Epub 2013 Oct 16. PMID 24129363